CLINICAL TRIAL: NCT00949754
Title: A Multi-Center, Randomized, Double Blind, Active-Controlled, Parallel Group Clinical Study to Evaluate the Dose Effect of Intradermal Injections of Apitox vs. Histamine in Subjects With Osteoarthritis Symptoms of the Knee
Brief Title: Apitox, Honeybee Venom Treatment for Osteoarthritis Pain and Inflammation
Acronym: HBV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apimeds, Inc. (Industry)
Responsible Party: Robert Brooks PhD, Chief Operating Officer US, Apimeds, Inc.
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: API092
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: honeybee venom; osteoarthritis; pain; knees
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Bee Venoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- histamine (Active Comparator): histamine in saline administered ID as active control for Apitox
  Interventions: Drug: honeybee venom (Apitoxin (Korea) Apitox (USA))
- Apitox pure honeybee venom (Experimental): ID study drug
  Interventions: Drug: honeybee venom (Apitoxin (Korea) Apitox (USA))

INTERVENTIONS:
Drug: honeybee venom (Apitoxin (Korea) Apitox (USA)) — multiple intradermal injections of 100 ug pure honeybee venom
  Other Names: Apitoxin (Korea) Apitox (USA)

SUMMARY:
The study will evaluate Apitox, pure honeybee venom as a treatment for pain and inflammation of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of one or both knees
* on stable NSAID or none due to intolerance
* women either post menopausal or on stable birth control
* no clinically significant disease or or abnormal laboratory values
* signed informed consent, communicate effectively, understand and comply with all study requirements

Exclusion Criteria:

* serious or unstable medical or psychological condition
* known sensitivity to honeybee venom, histamine or lidocaine
* history of asthma
* any clinically significant ECG abnormalities
* any clinically significant laboratory values OOR
* history of drug or alcohol abuse
* history of joint injury and forms of inflammatory arthritis

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
WOMAC | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher MH Kim, M.D., Study Chair — Apimeds, CEO; Robert Brooks, PhD, Study Director — Apimeds, Inc, US Chief Operating Officer
Locations (4):
- United States (4):
  - Radiant Research Inc., Pinellas Park, Florida
  - Radiant Research - Chicago, Chicago, Illinois
  - Radiant Research - Columbus, Columbus, Ohio
  - Radiant Research - San Antonio, San Antonio, Texas